CLINICAL TRIAL: NCT01689844
Title: Five Plus Nuts and Beans Trial
Brief Title: Randomized Trial of Tailored Dietary Advice to Lower Blood Pressure
Acronym: FivePlus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Edgar R. Miller, III, Principal Investigator, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NA00051935; P50CA148087-01 (Other Grant/Funding Number: National Heart, Lung, and Blood Institute)
Record Dates: First submitted 2012-04-27; First posted 2012-09-21 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: High Blood Pressure
Keywords: controlled high blood pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Behavioral, DASH Plus - Dietary advice (Active Comparator): This group will receive DASH diet advice and guided ordering of fruits, vegetables, nuts and beans that are high in potassium from a local supermarket.
  Interventions: Behavioral: DASH Plus
- DASH - C (Other): DASH C Group will receive brief DASH diet advice and will be able to make non- guided purchases of food products from the local supermarket.
  Interventions: Behavioral: DASH - C

INTERVENTIONS:
Behavioral: DASH Plus — DASH diet advice and guided shopping for high postassium foods at a local supermarket
  Arms: Behavioral, DASH Plus - Dietary advice
Behavioral: DASH - C — Brief DASH dietary advice, No shopping guidance at the local supermarket.
  Arms: DASH - C

SUMMARY:
The Five Plus Nuts & Beans Study is a randomized, controlled trial to compare two strategies for translating the results of the DASH (Dietary Approaches to Stop Hypertension) Study into practice for 120 African American participants who are on stable doses of antihypertensive medications. The first arm of our study offers minimal DASH-oriented dietary advice along with a food credit at a local supermarket where they make their own decision of what to eat. The second arm consists of a single one-hour session with a nutrition expert who provides choices and places an on-line order from a community grocery store (Santoni's Market) with targeted purchases of fruits, vegetables, nuts and beans. Our primary outcome is change in blood pressure at 8 weeks. Secondary outcomes are effects on glucose, uric acid, urine potassium excretion, and self-report consumption of fruits and vegetables during the same period.

DETAILED DESCRIPTION:
Unhealthy diets have many social determinants; however, there is a markedly lower availability of components of the DASH diet-recommended foods (such as fresh fruits and vegetables, skim milk and whole grain foods) in predominantly African-American and lower-income neighborhoods compared with Caucasian and higher-income neighborhoods. Unhealthy dietary consumption patterns contribute, in part, to hypertension through deficiencies in potassium, magnesium and vitamin C - all micronutrients with independent blood pressure-lowering effects. Furthermore, use of thiazide-based antihypertensive therapy often worsens deficiencies through increased urinary excretion. Strategies that take into account the multi-level nature of the problem of poor nutrition among low income African Americans are needed to improve adherence to dietary recommendations and reverse micronutrient deficiencies in hypertensive adults. The Five Plus Nuts & Beans Study is a randomized, controlled trial to compare two strategies for translating the results of the DASH (Dietary Approaches to Stop Hypertension) Study into practice for 120 African American participants who are on stable doses of antihypertensive medications. The first arm of our study offers minimal DASH-oriented dietary advice along with a food credit at a local supermarket where they make their own decision of what to eat. The second arm consists of a single one-hour session with a nutrition expert who provides choices and places an on-line order from a community grocery store (Santoni's Market) with targeted purchases of fruits, vegetables, nuts and beans. Following the initial contact, there is a weekly call with the coordinator for a $30 per week food delivery. Food orders are delivered for pick-up weekly by participants at a Baltimore Public Library in participant's neighborhood. Our primary outcome is change in blood pressure at 8 weeks. Secondary outcomes are effects on glucose, uric acid, urine potassium excretion, and self-report consumption of fruits and vegetables during the same period. After completion of the active phase of the trial, we will follow blood pressures in the electronic medical record for one year to assess long-term effects.

ELIGIBILITY:
Inclusion Criteria:

* must be age 21 or older,
* have a diagnosis of hypertension or pre-hypertension
* under regular care with their physician, and
* compliant with medications.
* systolic blood pressure of 120-140 mmHg and/or
* a diastolic blood pressure of 80-90 mmHg (average of two visits)
* on stable doses of antihypertensive medications for a minimum of two months prior to randomization, (and for the duration of the study).
* be able to follow all trial procedures.

Exclusion Criteria:

* cardiovascular event within 6 months,
* chronic disease that might interfere with trial participation (e.g. chronic kidney disease (estimated GFR < 60 cc/min),
* unwillingness or inability to adopt a DASH-like diet, and
* consumption of more than 14 alcoholic drinks per week,
* poorly controlled diabetes (Hemoglobin A1c >9%),
* use of insulin,
* use of mineral supplements or an unwillingness to stop supplements one month prior to randomization and refrain from the supplements during the study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2012-04; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | 8-wks follow-up
  Daytime systolic blood pressure determined by OMRON 907-xl blood pressure monitoring, will be the primary outcome measurement

SECONDARY OUTCOMES:
Fasting glucose, lipids and uric acid; urine K and Na excretion | 8-wks follow-up
  Fasting blood collections will occur in the morning after an overnight fast.

CONTACTS AND LOCATIONS:
Overall Officials: Edgar R Miller III, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Community Physicians, East Baltimore Medical Center, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Juraschek SP, White K, Tang O, Yeh HC, Cooper LA, Miller ER 3rd. Effects of a Dietary Approach to Stop Hypertension (DASH) Diet Intervention on Serum Uric Acid in African Americans With Hypertension. Arthritis Care Res (Hoboken). 2018 Oct;70(10):1509-1516. doi: 10.1002/acr.23515. Epub 2018 Aug 21. PMID 29342506